CLINICAL TRIAL: NCT05798650
Title: the Effect of Viewing Idealized Smile Images Versus Nature Images Via Social Media on Immediate Facial Satisfaction in Young Adults: a Randomized Controlled Trial.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr Maria Shakoor, Associate Professor, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: AIDM/ERC/11/2022/O1
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Facial Satisfaction
Keywords: facial satisfaction, ideal smile, nature, social media

STUDY DESIGN:
Intervention Model Description: After obtaining a written informed consent participants were divided into two groups, the experimental group and the control group. The experimental group had 60 Instagram user images of attractive smiles and the control group had 60 appearance- neutral Instagram images of nature.
  The neutral images for the control group were chosen with a hashtag nature on Instagram. These images only had nature and no people in them.
  A questionnaire was designed to investigate the effect of social networking site on facial and smile dissatisfaction, face related discrepancy and whether these effects differ from the use of appearance-neutral Instagram images. The questionnaire also assessed the use of social media and its effect on people.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instagram user images of attractive smiles (Experimental): the experimental group had 60 instagram user images of attractive smiles. The first author shortlisted 100 pictures with a hashtag #smile from Instagram. The photographs were of people with full attractive smile and well aligned teeth. These pictures were chosen from public profiles on Instagram. The photographs had an equal proportion of celebrity and non-celebrity faces and the age group was also similar to the people participating in the study (18-35 years).
  Interventions: Behavioral: facial dissatisfaction
- instagram images of nature (Placebo Comparator): the control group had 60 appearance- neutral Instagram images of nature. The neutral images for the control group were chosen with a hashtag nature on Instagram. These images only had nature and no people in them.
  Interventions: Behavioral: facial dissatisfaction

INTERVENTIONS:
Behavioral: facial dissatisfaction — Facial dissatisfaction was measured using orofacial aesthetic scale. Participants were asked about how they feel about their smile at that point of time.
  The state appearance comparison scale was used to see what the participants thought about their own appearance, their comparison to photographs, and the comparison of their smile, teeth and face to the photographs.
  Other Names: state appearance comaprison

SUMMARY:
The study was conducted to investigate the effect of social networking site on facial and smile dissatisfaction, face related discrepancy, and whether these effects differ from the use of appearance-neutral Instagram images.

DETAILED DESCRIPTION:
The study was conducted to investigate the effect of social networking site on facial and smile dissatisfaction, face related discrepancy, and whether these effects differ from the use of appearance-neutral Instagram images.

A simple random sampling technique was used for the recruitment of participants in this technique. Participants were both male and female undergraduate and graduate students. The participants were told that it is a study on social media. Participants were 18-35 years as 90% of Instagram users are aged between 18-35 years. Two sets of images were compiled for this study. One set had Instagram user images of attractive smiles. The other set had appearance-neutral Instagram images of nature. All the images were chosen from public Instagram images.

The first author shortlisted 100 pictures with a hashtag #smile from Instagram. The photographs were of people with full attractive smile and well aligned teeth. These pictures were chosen from public profiles on Instagram. The photographs had an equal proportion of celebrity and non-celebrity faces and the age group was also similar to the people participating in the study (18-35 years).

The neutral images for the control group were chosen with a hashtag nature on Instagram. These images only had nature and no people in them.

The stimulus material were chosen from Instagram. The images were tested by using a 5 point Likert scale by a team with 3 members, an orthodontist, a prosthodontist and a restorative dentist. The images were judged by the attractiveness of smile and teeth (1=very attractive, 5=very unattractive), image quality (1=very good quality, 5=not good quality), general appeal (1=very appealing, 5=not at all appealing) and enjoyment (1=very enjoyable, 2=not at all enjoyable). Out of 100 images, total 60 will be selected.

After obtaining a written informed consent participants were divided into two groups, the experimental group and the control group. The experimental group will view 60 images of attractive smiles on their phone and the control group will view 60 appearance- neutral Instagram images of nature.

A questionnaire was designed to investigate the effect of social networking site on facial and smile dissatisfaction, face related discrepancy and whether these effects differ from the use of appearance-neutral Instagram images. The questionnaire also assessed the use of social media and its effect on people.

The questionnaire consisted of general information including name, age and gender. The participants were also asked about their history of orthodontic / aesthetic / psychological treatments.

Facial dissatisfaction was measured using orofacial aesthetic scale and smile aesthetic satisfaction scale. Participants were asked about how they feel about their smile at that point of time. Answer was assessed using visual analogue scale. Further the participants were asked about their level of satisfaction with their smile using 3 point Likert scale.

The state appearance comparison scale was used to see what the participants thought about their own appearance, their comparison to photographs, and the comparison of their smile, teeth and face to the photographs. This was assessed using a 7 point Likert scale.

The state variant of self-discrepancy index was used to measure appearance discrepancy. Participants were asked about 5 things they would like to change in their appearance based on their facial and dental aesthetics.

the participants were also asked about their number of followers on Instagram, the number of personal friends they follow on Instagram, the number of celebrities they follow on Instagram.

ELIGIBILITY:
Inclusion Criteria:

* college graduates
* User of one social networking site (Instagram)

Exclusion Criteria:

* low socioeconomic status
* user of social networking sites other then instagram.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
the effect of viewing idealized smile images vs nature images via social media on immediate facial satisfaction. | 5 minutes
  The study was conducted to investigate the effect of social networking site on facial and smile dissatisfaction, face related discrepancy, and whether these effects differ from the use of appearance-neutral Instagram images.

CONTACTS AND LOCATIONS:
Overall Officials: dr maria shakoor, bds,fcps, Principal Investigator — Altamash Institute of Dental Medicine
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan